CLINICAL TRIAL: NCT01337050
Title: A Phase I Pharmacokinetic And Pharmacodynamic Study Of Pf-03446962 In Asian Patient With Advanced Solid Tumors
Brief Title: Asian Phase I Study Of PF-03446962
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: A8471004
Record Dates: First submitted 2011-04-06; First posted 2011-04-18 (Estimated); Results first posted 2015-08-28 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Neoplasms
Keywords: Hepatocellular Carcinoma; Advanced/Metastatic solid tumors
MeSH Terms: conditions — Neoplasms; Carcinoma, Hepatocellular | interventions — ascrinvacumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): PF-03446962
  Interventions: Drug: PF-03446962

INTERVENTIONS:
Drug: PF-03446962 — PF 03446962 given by a 1 hour IV infusion. Each patient will initially receive the first dose on Cycle 1 Day 1 with a 28 day observation period. Cycle 2 will start on Day 29. The dosing interval will be 14 days for Cycle 2 and subsequent cycles.

SUMMARY:
This is an Asian Phase 1, multi center, open label, single arm study of PF 03446962 with dose escalation and designed to define the Maximum Tolerated Dose [MTD] and the Recommended Phase 2 Dose [RP2D].

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of stomach cancer
* advanced/metastasis solid tumor refractory or intolerant to established therapy
* adequate blood chemistry, blood counts and kidney/liver function
* willing to participate to study requirements and sign an informed consent document

Exclusion Criteria:

* Chemotherapy, radiotherapy, or any investigational cancer therapy within 4 weeks of first dose of study medication
* excessive toxicities related to prior therapies
* pregnant or breastfeeding patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-07; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- National Cancer Center Hospital East, Kashiwa, Chiba, Japan
- Seoul National University Hospital/Department of Internal Medicine, Seoul, South Korea

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8471004&StudyName=Asian%20Phase%20I%20Study%20Of%20PF-03446962

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-03446962 4.5 mg/kg: PF-03446962 4.5 milligram per kilogram (mg/kg) intravenous infusion over 1 hour on Day 1 of each cycle. Cycle 1 was of 28 days duration and all subsequent cycles were of 14 days duration.
- PF-03446962 7.0 mg/kg: PF-03446962 7.0 mg/kg intravenous infusion over 1 hour on Day 1 of each cycle. Cycle 1 was of 28 days duration and all subsequent cycles were of 14 days duration.
- PF-03446962 10.0 mg/kg: PF-03446962 10.0 mg/kg intravenous infusion over 1 hour on Day 1 of each cycle. Cycle 1 was of 28 days duration and all subsequent cycles were of 14 days duration.
Period: Overall Study
Arm/Group | PF-03446962 4.5 mg/kg | PF-03446962 7.0 mg/kg | PF-03446962 10.0 mg/kg
Started | 4 | 13 | 19
Completed | 0 | 0 | 0
Not Completed | 4 | 13 | 19
Not completed — Death | 0 | 0 | 4
Not completed — Other | 4 | 6 | 8
Not completed — Participants refused further follow-up | 0 | 7 | 7

BASELINE CHARACTERISTICS:
Population: Full analysis set included all enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-03446962 4.5 mg/kg | PF-03446962 7.0 mg/kg | PF-03446962 10.0 mg/kg | Total
Number analyzed (Participants) | 4 | 13 | 19 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (10.9) | 56.5 (12.4) | 57.7 (13.1) | 57.4 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 5 | 11
  Male | 3 | 8 | 14 | 25

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: The MTD was defined as the highest dose of PF-03446962 associated with the occurrence of Dose Limiting Toxicities (DLTs) in at most 1 of 6 participants with the next higher dose having at least 2/3 or 2/6 participants experiencing DLTs (that is (i.e.) Maximum Administrated Dose). DLT is defined if the participants meets the following criteria during the first 6 weeks of treatment, possibly attributable to PF-03446962. Neutropenia grade 4 (less than [< ])500/cubic millimeter [mm^ 3]) lasting for greater than equal to (>=) 8 days; Febrile Neutropenia >= Grade 3; Neutropenic Infection >= Grade 3; Grade 4 thrombocytopenia (<25,000/mm^3); Grade 3 thrombocytopenia (<50,000/mm^3) with active bleeding; Grade 3 or higher non-hematological toxicity.
Time Frame: Baseline up to Week 6
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study medication. Here "N" (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Number; unit: mg/kg
Groups:
- PF-03446962: PF-03446962 4.5, 7.0 or 10.0 mg/kg intravenous infusion over 1 hour on Day 1 of each cycle. Cycle 1 was of 28 days duration and all subsequent cycles were of 14 days duration.
Arm/Group | PF-03446962
Number analyzed (Participants) | 12
mg/kg | 10.0

2. Primary Outcome: Recommended Phase-2 Dose (RP2D)
Description: RP2D was determined by a comprehensive assessments based on all the safety data, efficacy data, pharmacokinetics profile and biomarker data using blood and tumor samples.
Time Frame: Baseline up to 28 days after last dose of study medication
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study medication.
Measure: Number; unit: mg/kg
Arm/Group | PF-03446962
Number analyzed (Participants) | 36
mg/kg | 7.0

3. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pre-treatment state. AEs included both SAEs and non-serious adverse events (non-SAEs).
Time Frame: Baseline up to 28 days after last dose
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-03446962 4.5 mg/kg | PF-03446962 7.0 mg/kg | PF-03446962 10.0 mg/kg
Number analyzed (Participants) | 4 | 13 | 19
participants
  AEs | 3 | 13 | 19
  SAEs | 0 | 1 | 1

4. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) Based on Severity
Description: Adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. AE was assessed according to severity; Grade 1 (Mild Adverse Event), Grade 2 (Moderate Adverse Event), Grade 3 (Severe Adverse Event), Grade 4 (Life- Threatening or Disabling Adverse Event), Grade 5 (Death Related to Adverse Event).
Time Frame: Baseline up to 28 days after last dose
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-03446962 4.5 mg/kg | PF-03446962 7.0 mg/kg | PF-03446962 10.0 mg/kg
Number analyzed (Participants) | 4 | 13 | 19
participants
  Grade 1 | 0 | 4 | 5
  Grade 2 | 1 | 3 | 6
  Grade 3 | 2 | 4 | 8
  Grade 4 | 0 | 1 | 0
  Grade 5 | 0 | 1 | 0

5. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both SAEs and non-serious adverse events (non-SAEs). Relatedness to study drug was assessed based on investigator's discretion.
Time Frame: Baseline up to 28 days after last dose
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-03446962 4.5 mg/kg | PF-03446962 7.0 mg/kg | PF-03446962 10.0 mg/kg
Number analyzed (Participants) | 4 | 13 | 19
participants
  AEs | 3 | 9 | 14
  SAEs | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Laboratory Abnormalities
Description: Laboratory abnormalities were segregated into hematology, chemistry, coagulation and urinalysis test. It had been graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) into Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe) and Grade 4 (Life-threatening). Participants with abnormality of any of these grades are reported.
Time Frame: Baseline up to 28 days after last dose
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-03446962 4.5 mg/kg | PF-03446962 7.0 mg/kg | PF-03446962 10.0 mg/kg
Number analyzed (Participants) | 4 | 13 | 19
participants
  Anemia | 2 | 10 | 13
  Hemoglobin increased | 1 | 1 | 1
  Lymphocyte count increased | 0 | 2 | 2
  Lymphopenia | 2 | 1 | 5
  Neutrophils (absolute) | 0 | 1 | 1
  Platelets | 0 | 5 | 11
  White Blood Cells (WBC) | 1 | 2 | 1
  Alanine aminotransferase (ALT) | 2 | 5 | 9
  Alkaline phosphatase | 2 | 7 | 13
  Amylase | 1 | 3 | 5
  Aspartate aminotransferase (AST) | 1 | 8 | 13
  Total bilirubin | 0 | 4 | 4
  Creatinine | 4 | 13 | 18
  Hypercalcemia | 0 | 1 | 2
  Hyperglycemia | 4 | 13 | 17
  Hyperkalemia | 1 | 2 | 4
  Hypernatremia | 0 | 0 | 0
  Hypoalbuminemia | 3 | 6 | 10
  Hypocalcemia | 2 | 5 | 5
  Hyponatremia | 3 | 4 | 7
  Hypophosphatemia | 1 | 3 | 5
  Lipase | 0 | 7 | 2
  Prothrombin time (PT) | 1 | 4 | 7
  PT International Normalized Ratio(INR) | 1 | 2 | 3
  Urine protein | 4 | 10 | 11
  Hypoglycemia | 0 | 1 | 0

7. Secondary Outcome: Maximum Observed Serum Concentration (Cmax)
Time Frame: 0 (pre dose), 0.5, 1 (right before the end of infusion), 1.5, 2, 5, 8, 24 hours after the start of infusion of the first dose on Day 1; Day 3, 5, 8, 11, 15, 22 of Cycle 1
Population: Pharmacokinetic (PK) parameter analysis population included all participants treated who had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF-03446962 4.5 mg/kg | PF-03446962 7.0 mg/kg | PF-03446962 10.0 mg/kg
Number analyzed (Participants) | 4 | 13 | 19
nanogram per milliliter (ng/mL) | 89420 (47) | 121100 (34) | 169000 (28)

8. Secondary Outcome: Minimum Observed Serum Trough Concentration (Cmin)
Time Frame: as for outcome 7
Population: PK parameter analysis population included all participants treated who had at least 1 of the PK parameters of interest. Here "N" (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-03446962 4.5 mg/kg | PF-03446962 7.0 mg/kg | PF-03446962 10.0 mg/kg
Number analyzed (Participants) | 3 | 12 | 14
ng/mL | 6689 (47) | 14680 (22) | 22940 (27)

9. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: as for outcome 7
Population: PK parameter analysis population included all participants treated who had at least 1 of the PK parameters of interest.
Measure: Median (Full Range); unit: hours (hr)
Arm/Group | PF-03446962 4.5 mg/kg | PF-03446962 7.0 mg/kg | PF-03446962 10.0 mg/kg
Number analyzed (Participants) | 4 | 13 | 19
hours (hr) | 1.74 (47) [0.983 to 8.00] | 2.00 (22) [0.900 to 8.02] | 1.50 (27) [0.950 to 8.07]

10. Secondary Outcome: Area Under the Curve From Time Zero to 28 Days [AUC (0-28)]
Description: AUC (0-28)= Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-28).
Time Frame: as for outcome 7
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | PF-03446962 4.5 mg/kg | PF-03446962 7.0 mg/kg | PF-03446962 10.0 mg/kg
Number analyzed (Participants) | 4 | 12 | 14
nanogram*hour per milliliter (ng*hr/mL) | 12360000 (36) | 21980000 (14) | 30360000 (22)

11. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast)
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast) for drug.
Time Frame: as for outcome 7
Population: PK parameter analysis population included all participants treated who had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-03446962 4.5 mg/kg | PF-03446962 7.0 mg/kg | PF-03446962 10.0 mg/kg
Number analyzed (Participants) | 4 | 13 | 19
ng*hr/mL | 12050000 (39) | 20500000 (30) | 26070000 (62)

12. Secondary Outcome: Systemic Clearance (CL)
Description: CL is a quantitative measure of the rate at which a drug substance is removed from the body.
Time Frame: as for outcome 7
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/hr)
Arm/Group | PF-03446962 4.5 mg/kg | PF-03446962 7.0 mg/kg | PF-03446962 10.0 mg/kg
Number analyzed (Participants) | 4 | 7 | 2
liter per hour (L/hr) | 0.01880 (31) | 0.01482 (20) | NA (NA) — Data was not reported if less than 3 participants data was available, as planned.

13. Secondary Outcome: Volume of Distribution (Vd)
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug.
Time Frame: as for outcome 7
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter (L)
Arm/Group | PF-03446962 4.5 mg/kg | PF-03446962 7.0 mg/kg | PF-03446962 10.0 mg/kg
Number analyzed (Participants) | 4 | 7 | 2
liter (L) | 7.535 (23) | 6.556 (23) | NA (NA) — Data was not analyzed if less than 3 participants were evaluable for the measure, as per planned analysis.

14. Secondary Outcome: Plasma Decay Half-Life (t1/2)
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 7
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: days
Arm/Group | PF-03446962 4.5 mg/kg | PF-03446962 7.0 mg/kg | PF-03446962 10.0 mg/kg
Number analyzed (Participants) | 4 | 7 | 2
days | 14.58 (2.2081) | 14.16 (1.7822) | NA (NA) — Data was not analyzed if less than 3 participants were evaluable for the measure, as per planned analysis.

15. Secondary Outcome: Soluble Proteins Level
Description: Soluble proteins related to Activin Receptor-Like Kinase 1 (ALK-1) signaling and angiogenesis signaling including Vascular adhesion molecule (VAM), Monocyte chemotactic protein 1 (MCP-1), Angiopoietin 2, Tear intercellular adhesive molecule 1 (ICAM-1), Soluble intracellular adhesion molecule 1 (SIAM-1), Soluble vascular adhesion molecule 1 (SVAM-1), Vascular endothelial growth factor A (VEGF-A), Vascular endothelial growth factor C (VEGF-C), Vascular endothelial growth factor D (VEGF-D), Soluble vascular endothelial growth factor- Receptor 1 (REC 1) (SVEGF-REC 1), Soluble vascular endothelial growth factor- REC 2 (SVEGF-REC 2), Soluble vascular endothelial growth factor- REC 3 (SVEGF-REC 3), Bone morphogenetic protein-9 (BMP-9), Endoglin, Transforming growth factor- beta 1 (TGF- Beta 1), Placental growth factor (PGF) was evaluated.
Time Frame: Baseline, Day 1, 0 hour (H), 6 H Cycle 1 Day 1, Day 22 of Cycle 1, Day 1 Cycle 2, Day 1 Cycle 3 and end of treatment (up to cycle 30)
Population: Biomarker analysis population included all enrolled and treated participants with baseline and on-treatment biomarker sample analyzed. Here "n"= participants who were evaluable for specified biomarker at given time point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: picogram per milliliter (pg/mL)
Arm/Group | PF-03446962 4.5 mg/kg | PF-03446962 7.0 mg/kg | PF-03446962 10.0 mg/kg
Number analyzed (Participants) | 4 | 13 | 19
picogram per milliliter (pg/mL)
  VAM: Baseline (n=0,1,10) | NA (NA) — Data was not available as no participant was evaluable. | 5769662.5 (NA) — Standard deviation could not be calculated because only 1 participant was evaluable. | 4529407.4 (2147607.09)
  VAM: Cycle1/Day1 0H(n=0,1,10) | NA (NA) — Data was not available as no participant was evaluable. | 5013301.1 (NA) — Standard deviation could not be calculated because only 1 participant was evaluable. | 4834240.9 (4649500.22)
  VAM: Cycle1/Day1 6H (n=0,1,10) | NA (NA) — Data was not available as no participant was evaluable. | 6403610.0 (NA) — Standard deviation could not be calculated because only 1 participant was evaluable. | 5787177.6 (4880400.90)
  VAM: Cycle1/Day22 (n=0,0,10) | NA (NA) — Data was not available as no participant was evaluable. | NA (NA) — Data was not available as no participant was evaluable. | 6388997.9 (3326806.56)
  VAM: Cycle2/Day1 (n=0,0,8) | NA (NA) — Data was not available as no participant was evaluable. | NA (NA) — Data was not available as no participant was evaluable. | 8156950.3 (8059603.45)
  VAM: Cycle3/Day1 (n=0,1,3) | NA (NA) — Data was not available as no participant was evaluable. | 3539105.4 (NA) — Standard deviation could not be calculated because only 1 participant was evaluable. | 6601473.2 (3524102.00)
  VAM: End of Treatment (n=0,3,5) | NA (NA) — Data was not available as no participant was evaluable. | 10329091.1 (1748797.03) | 5648426.5 (1095588.29)
  MCP-1: Baseline (n=4,13,19) | 1049.6 (202.58) | 934.8 (444.61) | 1016.7 (341.58)
  MCP-1: Cycle1/Day1 0H (n=4,13,19) | 916.9 (79.30) | 911.2 (233.53) | 867.9 (345.20)
  MCP-1: Cycle1/Day1 6H (n=4,13,19) | 1246.8 (453.48) | 1774.5 (1150.89) | 2283.8 (1462.53)
  MCP-1: Cycle1/Day22 (n=4,12,16) | 932.2 (241.45) | 870.5 (233.82) | 1201.5 (654.63)
  MCP-1: Cycle2/Day1 (n=3,12,14) | 1202.9 (208.51) | 864.1 (188.86) | 1154.6 (741.31)
  MCP-1: Cycle3/Day1 (n=2,8,5) | 857.5 (95.32) | 916.8 (288.98) | 797.8 (403.62)
  MCP-1: End of Treatment (n=4,7,11) | 811.3 (185.47) | 1066.0 (451.04) | 1144.0 (547.92)
  Angioprotein-2: Baseline (n=4,13,19) | 358.7 (183.72) | 490.5 (300.64) | 730.1 (800.18)
  Angioprotein-2: Cycle1/Day1 0H (n=4,13,19) | 369.9 (167.24) | 439.2 (190.70) | 654.3 (686.73)
  Angioprotein-2: Cycle1/Day1 6H (n=4,13,19) | 282.1 (130.38) | 416.0 (239.46) | 792.7 (813.77)
  Angioprotein-2: Cycle1/Day22 (n=4,12,16) | 406.8 (234.83) | 503.4 (242.67) | 1282.8 (1901.84)
  Angioprotein-2: Cycle2/Day1 (n=3,12,14) | 269.5 (122.91) | 513.6 (280.22) | 752.2 (568.44)
  Angioprotein-2: Cycle3/Day1 (n=2,8,5) | 309.1 (48.30) | 510.8 (256.27) | 416.4 (514.40)
  Angioprotein-2: End of Treatment (n=4,7,11) | 288.6 (154.63) | 666.1 (510.48) | 1147.2 (1452.48)
  ICAM-1: Baseline (n=0,1,10) | NA (NA) — Data was not available as no participant was evaluable. | 1277073.8 (NA) — Standard deviation could not be calculated because only 1 participant was evaluable. | 931954.7 (1058110.51)
  ICAM-1: Cycle1/Day1 0H (n=0,1,10) | NA (NA) — Data was not available as no participant was evaluable. | 878849.0 (NA) — Standard deviation could not be calculated because only 1 participant was evaluable. | 844534.8 (802742.55)
  ICAM-1: Cycle1/Day1 6H (n=0,1,10,) | NA (NA) — Data was not available as no participant was evaluable. | 806572.4 (NA) — Standard deviation could not be calculated because only 1 participant was evaluable. | 915166.4 (923611.09)
  ICAM-1: Cycle1/Day22(n=0,0,10) | NA (NA) — Data was not available as no participant was evaluable. | NA (NA) — Data was not available as no participant was evaluable. | 1226089.9 (1128415.32)
  ICAM-1: Cycle2/Day1 (n=0,0,8) | NA (NA) — Data was not available as no participant was evaluable. | NA (NA) — Data was not available as no participant was evaluable. | 827621.8 (367125.98)
  ICAM-1: Cycle3/Day1 (n=0,1,3) | NA (NA) — Data was not available as no participant was evaluable. | 479439.4 (NA) — Standard deviation could not be calculated because only 1 participant was evaluable. | 542607.5 (150328.01)
  ICAM-1: End of Treatment (n=0,3,5) | NA (NA) — Data was not available as no participant was evaluable. | 1271075.6 (515605.73) | 1651061.8 (2042387.17)
  SIAM-1: Baseline (n=4,12,9) | 701303.4 (294804.13) | 466302.8 (309842.34) | 525958.2 (113283.77)
  SIAM-1: Cycle1/Day1 0H (n=4,12,9) | 623840.0 (181192.64) | 504021.3 (256755.23) | 532390.8 (180640.87)
  SIAM-1: Cycle1/Day1 6H (n=4,12,9) | 604163.5 (214935.46) | 411628.1 (261009.28) | 569359.0 (201989.70)
  SIAM-1: Cycle1/Day22 (n=4,12,6) | 668593.1 (184915.57) | 501742.8 (320205.39) | 622325.0 (238791.57)
  SIAM-1: Cycle2/Day1 (n=3,12,6) | 552736.5 (184915.57) | 501742.8 (320205.39) | 622325.0 (238791.57)
  SIAM-1: Cycle3/Day1 (n=2,7,2) | 638075.4 (127112.48) | 598448.3 (317579.77) | 438595.7 (166268.03)
  SIAM-1: End of Treatment (n=4,4,6) | 628177.9 (163803.34) | 464669.7 (174245.04) | 719398.7 (231843.95)
  SVAM-1: Baseline (n=4,12,9) | 2135238.6 (849420.75) | 3651583.3 (2216213.70) | 2551024.9 (595975.01)
  SVAM-1: Cycle1/Day1 0H (n=4,12,9) | 2061387.9 (858687.41) | 3583328.2 (1998977.25) | 2620267.2 (1001526.82)
  SVAM-1: Cycle1/Day1 6H (n=4,12,9) | 2034173.6 (756983.20) | 3576192.6 (2751678.60) | 3071682.9 (1447507.40)
  SVAM-1: Cycle1/Day22 (n=4,12,6) | 2665272.7 (1159532.95) | 4276947.7 (2862681.78) | 3653830.7 (1746452.25)
  SVAM-1: Cycle2/Day1 (n=3,12,6) | 1892498.5 (68777.63) | 4628918.3 (3257637.40) | 3574717.1 (1661302.68)
  SVAM-1: Cycle3/Day1 (n=2,7,2) | 2117070.8 (747786.71) | 4755433.2 (2598745.99) | 2349177.5 (638957.67)
  SVAM-1: End of Treatment (n=4,4,6) | 3802384.0 (2865638.01) | 3318897.7 (1948986.96) | 3748602.8 (1332529.49)
  VEGF-A: Baseline (n=4,13,19) | 429.4 (208.76) | 889.8 (1475.25) | 463.4 (425.39)
  VEGF-A: Cycle1/Day1 0H (n=4,13,19) | 455.4 (175.23) | 595.3 (628.14) | 410.3 (419.93)
  VEGF-A: Cycle1/Day1 6H (n=4,13,19) | 438.6 (210.06) | 631.9 (644.09) | 460.5 (344.90)
  VEGF-A: Cycle1/Day22 (n=4,12,16) | 703.7 (416.74) | 462.8 (381.85) | 529.1 (511.82)
  VEGF-A: Cycle2/Day1 (n=3,12,14) | 941.0 (415.59) | 508.0 (406.78) | 524.7 (541.09)
  VEGF-A: Cycle3/Day1 (n=2,8,5) | 904.2 (1051.75) | 355.7 (259.00) | 373.5 (124.19)
  VEGF-A: End of Treatment (n=4,7,11) | 632.2 (676.85) | 491.6 (329.84) | 556.7 (740.20)
  VEGF-C: Baseline (n=4,13,19) | 110.6 (64.88) | 112.0 (91.80) | 139.9 (92.74)
  VEGF-C: Cycle1/Day1 0H (n=4,13,19) | 104.2 (62.45) | 98.2 (101.48) | 95.6 (81.09)
  VEGF-C: Cycle1/Day1 6H (n=4,13,19) | 81.8 (52.85) | 79.3 (64.75) | 104.2 (91.99)
  VEGF-C: Cycle1/Day22 (n=4,12,16) | 115.0 (67.41) | 94.2 (90.41) | 105.1 (92.55)
  VEGF-C: Cycle2/Day1 (n=3,12,14) | 91.6 (61.06) | 93.0 (106.58) | 93.7 (96.83)
  VEGF-C: Cycle3/Day1 (n=2,8,5) | 31.3 (0.00) | 82.2 (124.89) | 128.3 (116.64)
  VEGF-C: End of Treatment (n=4,7,11) | 70.9 (60.02) | 93.3 (111.24) | 64.7 (68.37)
  VEGF-D: Baseline (n=4,13,19) | 988.6 (208.49) | 1349.5 (1133.71) | 1176.4 (361.43)
  VEGF-D: Cycle1/Day1 0H (n=4,13,19) | 941.6 (114.91) | 1323.1 (962.53) | 1059.7 (365.10)
  VEGF-D: Cycle1/Day1 6H (n=4,13,19) | 881.9 (89.36) | 1341.9 (1154.09) | 1160.3 (389.49)
  VEGF-D: Cycle1/Day22 (n=4,12,16) | 853.9 (176.92) | 1327.6 (984.57) | 1365.8 (431.90)
  VEGF-D: Cycle2/Day1 (n=3,12,14) | 836.2 (161.42) | 1430.0 (1203.55) | 1315.8 (527.01)
  VEGF-D: Cycle3/Day1 (n=2,8,5) | 995.7 (263.82) | 1445.3 (1403.28) | 995.2 (443.14)
  VEGF-D: End of Treatment (n=4,7,11) | 809.4 (176.66) | 1494.1 (1000.50) | 1420.1 (402.57)
  SVEGF-REC 1: Baseline (n=4,13,19) | 152.3 (29.59) | 162.3 (60.10) | 228.5 (88.14)
  SVEGF-REC 1: Cycle1/Day1 0H (n=4,13,19) | 114.0 (51.72) | 1397.1 (4204.03) | 3196.4 (10603.61)
  SVEGF-REC 1: Cycle1/Day1 6H (n=4,13,19) | 116.9 (16.94) | 177.1 (81.20) | 255.2 (95.68)
  SVEGF-REC 1: Cycle1/Day22 (n=4,12,16) | 132.0 (39.82) | 170.9 (93.07) | 299.4 (138.60)
  SVEGF-REC 1: Cycle2/Day1 (n=3,12,14) | 447.4 (467.46) | 222.5 (142.78) | 261.0 (115.68)
  SVEGF-REC 1: Cycle3/Day1 (n=2,8,5) | 103.8 (29.27) | 155.5 (80.26) | 192.5 (82.80)
  SVEGF-REC 1: End of Treatment (n=4,7,11) | 113.7 (33.47) | 234.2 (172.30) | 276.8 (227.19)
  SVEGF-REC 2: Baseline (n=4,13,19) | 7436.6 (1857.86) | 6888.7 (2231.62) | 8440.8 (2437.27)
  SVEGF-REC 2: Cycle1/Day1 0H (n=4,13,19) | 7914.2 (2988.27) | 7026.7 (2025.46) | 7741.2 (2133.30)
  SVEGF-REC 2: Cycle1/Day1 6H (n=4,13,19) | 7870.7 (3373.09) | 6586.3 (2081.36) | 8378.4 (1904.55)
  SVEGF-REC 2: Cycle1/Day22 (n=4,12,16) | 7235.8 (2807.65) | 7069.1 (2453.67) | 8493.1 (1844.69)
  SVEGF-REC 2: Cycle2/Day1 (n=3,12,14) | 7597.3 (3168.18) | 7245.4 (2560.56) | 7965.4 (2421.06)
  SVEGF-REC 2: Cycle3/Day1 (n=2,8,5) | 8516.8 (3960.15) | 6827.8 (2613.39) | 8193.9 (2074.23)
  SVEGF-REC 2: End of Treatment (n=4,7,11) | 6714.4 (2171.59) | 6908.6 (2872.56) | 8963.3 (1366.42)
  SVEGF-REC 3: Baseline (n=4,13,19) | 456712.6 (63869.92) | 332957.5 (114561.87) | 434940.1 (109510.31)
  SVEGF-REC 3: Cycle1/Day1 0H (n=4,13,19) | 406786.4 (11524.53) | 355960.5 (132035.48) | 407148.7 (92393.49)
  SVEGF-REC 3: Cycle1/Day1 6H (n=4,13,19) | 395896.6 (61076.24) | 336962.5 (141091.61) | 416266.6 (90886.33)
  SVEGF-REC 3: Cycle1/Day22 (n=4,12,16) | 374514.7 (33518.13) | 310883.6 (87289.24) | 454274.1 (141305.28)
  SVEGF-REC 3: Cycle2/Day1 (n=3,12,14) | 405961.9 (34525.64) | 317659.8 (79198.45) | 450339.2 (162644.43)
  SVEGF-REC 3: Cycle3/Day1 (n=2,8,5) | 421505.5 (23124.80) | 289021.4 (73419.94) | 311026.0 (93213.81)
  SVEGF-REC 3: End of Treatment (n=4,7,11) | 345569.6 (19964.62) | 307319.1 (99790.00) | 434549.1 (95476.81)
  BMP-9: Baseline (n=4,13,19) | 8.3 (4.77) | 64.5 (155.34) | 24.8 (18.39)
  BMP-9: Cycle1/Day1 0H (n=4,13,19) | 7.4 (5.00) | 47.3 (114.00) | 22.0 (12.61)
  BMP-9: Cycle1/Day1 6H (n=4,13,19) | 16.7 (8.95) | 58.6 (130.87) | 33.4 (15.93)
  BMP-9: Cycle1/Day22 (n=4,12,16) | 8.9 (6.39) | 49.8 (121.48) | 25.7 (12.26)
  BMP-9: Cycle2/Day1 (n=3,12,14) | 8.1 (5.01) | 61.5 (158.39) | 24.7 (12.58)
  BMP-9: Cycle3/Day1 (n=2,8,5) | 16.5 (16.33) | 84.8 (194.91) | 25.2 (10.90)
  BMP-9: End of Treatment (n=4,7,11) | 11.2 (6.09) | 123.3 (259.17) | 47.0 (70.74)
  Endoglin: Baseline (n=4,13,19) | 22292.9 (7065.67) | 26312.5 (8345.99) | 31096.0 (7553.99)
  Endoglin: Cycle1/Day1 0H (n=4,13,19) | 21148.2 (4493.48) | 26514.1 (4171.10) | 29437.1 (8796.80)
  Endoglin: Cycle1/Day1 6H (n=4,13,19) | 20252.9 (3093.23) | 24385.0 (7947.74) | 29898.7 (7743.02)
  Endoglin: Cycle1/Day22 (n=4,12,16) | 20304.6 (3085.27) | 28106.4 (6786.70) | 39570.2 (11857.18)
  Endoglin: Cycle2/Day1 (n=3,12,14) | 18974.4 (2212.35) | 29533.7 (8065.27) | 35585.1 (8558.35)
  Endoglin: Cycle3/Day1 (n=2,8,5) | 20441.2 (5168.88) | 28063.4 (6794.28) | 33439.4 (7464.88)
  Endoglin: End of Treatment (n=4,7,11) | 21756.8 (5825.18) | 31653.3 (9829.63) | 33159.2 (10674.69)
  TGF-Beta1: Baseline (n=4,13,19) | 439154.4 (194384.01) | 288057.2 (95964.14) | 264779.6 (245081.23)
  TGF-Beta1: Cycle1/Day1 0H (n=4,13,19) | 420293.6 (154286.55) | 228313.8 (101963.47) | 187730.4 (173444.62)
  TGF-Beta1: Cycle1/Day1 6H (n=4,13,19) | 361727.2 (195371.45) | 240430.8 (97194.19) | 194814.7 (173849.07)
  TGF-Beta1: Cycle1/Day22 (n=4,12,16) | 322848.7 (122214.82) | 248764.0 (105171.95) | 169310.4 (187249.43)
  TGF-Beta1: Cycle2/Day1 (n=3,12,14) | 485627.2 (145104.03) | 253554.9 (97795.74) | 214255.5 (269963.90)
  TGF-Beta1: Cycle3/Day1 (n=2,8,5) | 355810.5 (308789.78) | 231920.2 (128882.61) | 280515.6 (270982.35)
  TGF-Beta1: End of Treatment (n=4,7,11) | 292378.4 (154058.94) | 235871.6 (129631.54) | 249663.6 (300797.29)
  PGF: Baseline (n=4,13,19) | 15.6 (16.56) | 10.7 (4.03) | 9.6 (4.80)
  PGF: Cycle1/Day1 0H (n=4,13,19) | 15.3 (13.03) | 12.7 (4.67) | 9.5 (4.40)
  PGF: Cycle1/Day1 6H (n=4,13,19) | 15.7 (9.90) | 14.8 (7.35) | 14.8 (7.29)
  PGF: Cycle1/Day22 (n=4,12,16) | 14.5 (8.19) | 9.6 (3.28) | 9.9 (6.58)
  PGF:Cycle2/Day1 (n=3,12,14) | 9.9 (1.25) | 10.1 (3.77) | 9.2 (5.15)
  PGF: Cycle3/Day1 (n=2,8,5) | 7.2 (0.28) | 8.2 (2.60) | 6.9 (1.87)
  PGF: End of Treatment (n=4,7,11) | 10.3 (8.28) | 7.9 (2.43) | 8.6 (5.15)

16. Secondary Outcome: Number of Participants With Human Anti-Human Antibody (HAHA)
Description: HAHA analysis was performed using validated, sensitive and specific chemiluminescence enzyme-linked immunosorbent assay (ELISA) methodology.
Time Frame: Baseline, Post-dose (Day 1 of every Cycle up to 28 days after last dose) up to Cycle 30
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-03446962 4.5 mg/kg | PF-03446962 7.0 mg/kg | PF-03446962 10.0 mg/kg
Number analyzed (Participants) | 4 | 13 | 19
participants
  Baseline | 0 (NA) | 1 (2147607.09) | 3 (2071432.82)
  Post-Dose | 0 (NA) | 0 (4649500.22) | 0 (4411233.60)

17. Secondary Outcome: Number of Participants With Best Overall Response (BOR)
Description: Number of participants with best overall response according to Response Evaluation Criteria in Solid Tumors (RECIST); Complete response (CR): disappearance of all lesions, Pathological lymph nodes' reduction in short axis (SA) to less than (<)10 millimeter (mm); Partial response (PR): greater than equal to (>=) 30% decrease in sum of longest dimensions (LD) of Target Lesions (TL) taking reference baseline sum LD; Progressive disease (PD):>=20% (>= 5 mm increase) increase sum of LD of TL taking as a reference smallest sum of LD recorded since treatment start, appearance of >=1 new lesions, unequivocal progression of existing non-TL, or appearance of >=1 new lesion; Stable disease (SD): insufficient shrinkage to qualify for PR, insufficient increase to qualify for PD taking reference smallest sum of the LD since treatment start. Confirmed response=that persist at least 4 weeks after initial documentation.
Time Frame: Baseline, thereafter every 6 weeks up to end of treatment (up to Cycle 30)
Population: Response evaluable population included all enrolled participants with measurable disease who received at least 1 dose of PF-03446962 and had an adequate baseline tumor assessment. Here "N" (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | PF-03446962 4.5 mg/kg | PF-03446962 7.0 mg/kg | PF-03446962 10.0 mg/kg
Number analyzed (Participants) | 4 | 13 | 18
participants
  CR | 0 (NA) | 0 (2147607.09) | 0 (2071432.82)
  PR | 0 (NA) | 0 (4649500.22) | 0 (4411233.60)
  SD | 1 (NA) | 4 (8059603.45) | 4 (8059603.45)
  PD | 2 (NA) | 7 (3524102.00) | 13 (3259456.10)
  Symptomatic Deterioration | 0 (1748797.03) | 0 (1095588.29) | 1 (2725448.88)
  Early Death | 0 | 1 | 0
  Indeterminate | 1 | 1 | 0

18. Secondary Outcome: Number of Participants With Clinical Benefit Response (CBR)
Description: Number of participant with clinical benefit response (CBR): CBR was defined as CR, PR, SD >12 weeks, SD<12weeks or PD according to RECIST criteria; Complete response (CR): disappearance of all lesions, Pathological lymph nodes' reduction in short axis (SA) to <10 mm; Partial response (PR): >=30% decrease in sum of longest dimensions (LD) of Target Lesions (TL) taking reference baseline sum LD; Progressive disease (PD):>=20% (>= 5 mm increase) increase sum of LD of TL taking as a reference smallest sum of LD recorded since treatment start, appearance of >=1 new lesions, unequivocal progression of existing non-TL, or appearance of >=1 new lesion; Stable disease (SD): insufficient shrinkage to qualify for PR, insufficient increase to qualify for PD taking reference smallest sum of the LD since treatment start.
Time Frame: Baseline, thereafter every 6 weeks up to end of treatment (up to Cycle 30)
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | PF-03446962 4.5 mg/kg | PF-03446962 7.0 mg/kg | PF-03446962 10.0 mg/kg
Number analyzed (Participants) | 4 | 13 | 18
participants | 1 | 4 | 4

19. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from the first dose of study treatment to the first documentation of objective tumor progression or to death due to any cause, whichever occurred first. PFS calculated as (Months) = (first event date minus randomization or the first dose date plus 1) divided by 30.44). PFS was calculated using the median, and 95% Confidence Intervals (CIs) and Progressive disease (PD):>=20% (>= 5 mm increase) increase sum of LD of TL taking as a reference smallest sum of LD recorded since treatment start, appearance of >=1 new lesions, unequivocal progression of existing non-TL, or appearance of >=1 new lesion.
Time Frame: Baseline, thereafter every 6 weeks up to end of treatment (up to Cycle 30)
Population: as for outcome 17
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PF-03446962 4.5 mg/kg | PF-03446962 7.0 mg/kg | PF-03446962 10.0 mg/kg
Number analyzed (Participants) | 4 | 13 | 18
months | 2.8 (NA) [1.2 to 2.9] | 1.8 (2147607.09) [1.3 to 5.6] | 1.3 (2071432.82) [1.2 to 1.5]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as non-serious in another subject, or one subject may have experienced both a serious and non-serious event during the study.
Arm/Group | PF-03446962 4.5 mg/kg | PF-03446962 7.0 mg/kg | PF-03446962 10.0 mg/kg
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/13 | 1/19
Other Adverse Events (participants affected / at risk) | 3/4 | 13/13 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-03446962 4.5 mg/kg (N=4) | PF-03446962 7.0 mg/kg (N=13) | PF-03446962 10.0 mg/kg (N=19)
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-03446962 4.5 mg/kg (N=4) | PF-03446962 7.0 mg/kg (N=13) | PF-03446962 10.0 mg/kg (N=19)
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 3
Conjunctival haemorrhage (Eye disorders) | 0 | 3 | 1
Eye pain (Eye disorders) | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 2
Anorectal disorder (Gastrointestinal disorders) | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2
Asthenia (General disorders) | 0 | 1 | 1
Chest pain (General disorders) | 0 | 1 | 0
Chills (General disorders) | 0 | 1 | 0
Face oedema (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 2 | 2
Injection site extravasation (General disorders) | 0 | 1 | 0
Oedema (General disorders) | 0 | 1 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 3 | 10
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1
Enteritis infectious (Infections and infestations) | 0 | 1 | 0
Pseudofolliculitis barbae (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 2
Viral infection (Infections and infestations) | 0 | 1 | 0
Eschar (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural site reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Amylase increased (Investigations) | 0 | 2 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 2
Blood albumin decreased (Investigations) | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 4
Blood bilirubin increased (Investigations) | 0 | 1 | 1
C-reactive protein increased (Investigations) | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 1 | 1
Haemoglobin decreased (Investigations) | 1 | 0 | 0
Lipase increased (Investigations) | 0 | 1 | 1
Lymphocyte count decreased (Investigations) | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 2 | 3
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Liver carcinoma ruptured (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 2 | 0
Headache (Nervous system disorders) | 0 | 0 | 3
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0
Monoplegia (Nervous system disorders) | 0 | 0 | 1
Nervous system disorder (Nervous system disorders) | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1
Atonic urinary bladder (Renal and urinary disorders) | 0 | 0 | 1
Azotaemia (Renal and urinary disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 1 | 1
Proteinuria (Renal and urinary disorders) | 2 | 2 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 | 3 | 0

LIMITATIONS AND CAVEATS:
Designation of primary and secondary endpoints was based on study team's inputs, as the endpoints were not prioritized in the study protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.